CLINICAL TRIAL: NCT01013675
Title: Randomized, Double-blind, Active -Controlled Trial to Assess Safety and Immunogenicity of Solvay's Cell-derived Influenza Vaccine, Including Revaccination, in Elderly Subjects
Brief Title: Immunogenicity and Safety of a Cell-derived Influenza Vaccine in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S203.2.009; 2009-014767-40 (EudraCT Number)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Influenza Vaccines
Keywords: influenza; active-controlled; Phase 2
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 15 mcg hemagglutinin (HA) per viral strain; 0.5 mL single dose
  Interventions: Biological: Influenza Vaccine
- 2 (Active Comparator): 15 mcg hemagglutinin (HA) per viral strain; 0.5 mL single dose
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in cell cultures
  Arms: 1
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in egg (influvac ®)
  Arms: 2

SUMMARY:
A controlled, double-blind study to determine the immunogenicity and safety of influenza cell derived vaccine in elderly subjects.

DETAILED DESCRIPTION:
This current phase II study is to pursue objectives similar to those of the ongoing adult phase II trial, but to expand into the elderly population who are more than 60 years of age. The results of this randomized, double blind, egg derived influenza vaccine (Influvac) - controlled, parallel-trial, in healthy elderly subjects are to be conducted over two consecutive years in multiple centers in Europe. At study initiation 600 subjects will be randomly allocated to receive the cell-derived or egg-derived influenza vaccine. At start of the second year subjects will be randomly re-allocated following stratification based upon the initial drug they were allocated and had received.

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to give informed consent and able to adhere to all protocol required study procedures.
2. Men and women (elderly)
3. Being in good health as judged by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria

1. Known to be allergic to constituents of the vaccine.
2. A serious adverse reaction after a previous (influenza) vaccination. Presence of any significant condition that may prohibit inclusion as determined by the investigator.
3. Having received vaccination against influenza or lab confirmed influenza within the previous six months before study vaccination.

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the immunogenicity of the cell-derived subunit vaccine three weeks after vaccination, by applying the CHMP criteria for immunogenicity. | 3 weeks
To assess the safety and tolerability of the cell-derived vaccine and compare to an egg-derived influenza vaccine. | 6 months
To assess the safety and tolerability of the cell-derived vaccine following revaccination. | 6 months

SECONDARY OUTCOMES:
To assess the immunogenicity of the cell-derived subunit vaccine three weeks after revaccination, by applying the CHMP criteria for immunogenicity. | 3 weeks
To assess the long-term immunogenicity (6 months) of the cell-derived subunit vaccine. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanka de Voogd, MD, Study Director — Abbott Healthcare Products B.V
Locations (12):
- Czechia (2):
  - Site Reference ID/Investigator# 45005, Benátky nad Jizerou
  - Site Reference ID/Investigator# 45004, Hradec Králové
- Estonia (5):
  - Site Reference ID/Investigator# 45007, Paide
  - Site Reference ID/Investigator# 45012, Saku
  - Site Reference ID/Investigator# 45009, Tallinn
  - Site Reference ID/Investigator# 45010, Tallinn
  - Site Reference ID/Investigator# 45013, Tartu
- Lithuania (5):
  - Site Reference ID/Investigator# 45017, Kaunas
  - Site Reference ID/Investigator# 45015, Kaunas
  - Site Reference ID/Investigator# 45016, Kaunas
  - Site Reference ID/Investigator# 45018, Kaunas
  - Site Reference ID/Investigator# 45019, Klaipėda